CLINICAL TRIAL: NCT00778336
Title: Peripheral Use of AngioJet Rheolytic Thrombectomy With Mid-Length Catheters
Brief Title: A Prospective Observational Registry of Peripheral Use of AngioJet Rheolytic Thrombectomy With Mid-Length Catheters
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PEARL
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Results first posted 2011-04-26 (Estimated); Last update posted 2014-10-17 (Estimated); Status verified 2014-10

CONDITIONS: Peripheral Vascular Diseases; Thrombosis; Venous Thrombosis
Keywords: Peripheral Thrombosis; DVT; Limb Ischemia; AV Access; AngioJet; Thrombectomy
MeSH Terms: conditions — Peripheral Vascular Diseases; Thrombosis; Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Limb Ischemia: Patients presenting with limb ischemia for treatment
- Deep Vein Thrombosis: Patients presenting with deep vein thrombosis for treatment
- Hemodialysis Access: Patients presenting with thrombosed hemodialysis access for treatment
- Other Thrombotic Conditions: Patients presenting with thrombosed conditions other than limb ischemia, deep vein thrombosis or thrombosed hemodialysis access for treatment.

SUMMARY:
This registry collects observational data about how mid-length AngioJet catheters (ie XPEEDIOR and DVX models) are used in routine clinical practice.

DETAILED DESCRIPTION:
The PEARL Registry collects real world data about mid-length AngioJet catheters to:

* Characterize usage patterns, treatment approaches, and targeted vessels
* Document treatment strategies, including specific techniques and concomitant therapies
* Collect outcome data during initial hospitalization and at a 3-month follow-up phone call or visit
* Evaluate the frequency of specific clinical events in relation to risk factors, diagnosis, and treatments provided
* Identify treatment strategies that may optimize procedural and clinical outcomes, to facilitate development of treatment guidelines
* Offer sites a valuable resource for tracking usage and performance of the AngioJet System at their institution

Information collected by the PEARL Registry is intended for educational and clinical research purposes only.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been treated with a mid-length AngioJet catheter(defined as 90-120 cm in length)
* Patient has provided appropriate authorization per institutional policy and procedure.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with peripheral thrombosis treated with a AngioJet mid-length catheter that is indicated for thrombosis removal.
Sampling Method: Non-Probability Sample
Enrollment: 452 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence R. Blitz, MD, Principal Investigator — Chilton Memorial Hospital, Pompton Plains, NJ; Robert Lookstein, MD, Principal Investigator — Mount Sinai School of Medicine, NYC, NY; Eugene Simoni, MD, Principal Investigator — Samaritan Vascular Institute, Dayton, OH

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting at a participating site who were clinically indicated for a peripheral interventional(venous or arterial) procedure with the mid-length (90cm or 120cm catheters) catheter were offered the opportunity to participate. Patients were recruited from January 2007 thru December 2009.
Groups:
- Limb Ischemia: Patients with limb ischemia treated with a midlength AngioJet catheter.
- Deep Vein Thrombosis: Patients with deep vein thrombosis treated with a midlength AngioJet catheter.
- Hemodialysis Access: Patients with thrombosed hemodialysis access treated with a midlength AngioJet catheter.
- Other Thrombotic Conditions: Patients with a thrombotic Condition other than limb ischemia, deep vein thrombosis or thrombosed hemodialysis access treated with a midlength AngioJet catheter.
Period: Index Procedure-Discharge
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Started | 198 | 170 | 72 | 12
Completed | 192 | 167 | 70 | 12
Not Completed | 6 | 3 | 2 | 0
Not completed — Death | 6 | 3 | 2 | 0
Period: 3 Month Follow Up
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Started | 192 | 167 | 70 | 12
Completed | 169 | 144 | 65 | 12
Not Completed | 23 | 23 | 5 | 0
Not completed — Lost to Follow-up | 15 | 20 | 3 | 0
Not completed — Death | 8 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions | Total
Number analyzed (Participants) | 198 | 170 | 72 | 12 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (14) | 52 (17) | 63 (13) | 63 (18) | 61 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88 | 64 | 34 | 6 | 192
  Male | 110 | 106 | 38 | 6 | 260
Region of Enrollment [Number; unit: participants]
  United States | 198 | 170 | 72 | 12 | 452

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Final Angiographic Results
Description: From the Index Procedure's Baseline (pre-endovascular treatment) and Final (post-endovascular treatment) angiograms,each vessel was assigned a value by the treating physician:
  1. complete occlusion (> 90% occlusion);
  2. substantial occlusion (50-90% occlusion OR <50% occlusion and >3cm in length);
  3. partial occlusion (<50% occlusion AND <3cm in length);
  4. patent (Without visable thrombus or occlusion).
  The levels of change (improvement) were calculated by subtracting the baseline assigned angiographic value from the final value.
Time Frame: Index Procedure ( pre-endovascular treatment and post-endovascular treatment)
Population: Intention to Treat (ITT)
Measure: Mean (Standard Error); unit: Occlusion Index
Groups:
- Limb Ischemia: Patients treated with a midlength Angiojet catheter for limb ischemia
- Deep Vein Thrombosis: Patients treated with a midlength Angiojet catheter for deep vein thrombosis
- Hemodialysis Access: Patients treated with a midlength Angiojet catheter for thrombosed hemodialysis access sites
- Other Thrombotic Conditions: Patients treated with a midlength Angiojet catheter for thrombotic conditions other than limb ischemia, deep vein thrombosis or thrombosed hemodialysis access
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Number analyzed (Participants) | 198 | 170 | 72 | 12
Occlusion Index
  Baseline (pre-treatment) Angiograph Value | 1.32 (0.04) | 1.37 (0.04) | 1.16 (0.05) | 1.89 (0.14)
  Final (post-treatment) Angiograph Value | 3.67 (0.05) | 3.67 (0.04) | 3.80 (0.07) | 3.54 (0.14)
  Levels of Change (baseline minus final values) | 2.36 (0.06) | 2.30 (0.05) | 2.63 (0.08) | 1.63 (0.18)
Statistical Analysis 1: Comparison: Limb Ischemia; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion > 0
Statistical Analysis 2: Comparison: Deep Vein Thrombosis; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion > 0
Statistical Analysis 3: Comparison: Hemodialysis Access; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion > 0
Statistical Analysis 4: Comparison: Other Thrombotic Conditions; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; Alternative hypothesis is change in occlusion > 0

2. Secondary Outcome: Rethrombosis
Description: The number of patients that had rethrombosed in the vessels treated during the index procedure (initial endovascular procedure).
Time Frame: 3 Month Follow Up
Measure: Number; unit: Participants
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Number analyzed (Participants) | 198 | 170 | 72 | 12
Participants | 17 | 11 | 14 | 0

3. Secondary Outcome: Description of Treatments by Thrombotic Condition
Description: The # of patients that were exposed to each treatment at least once in the given thrombotic condition.
Time Frame: Index Procedure
Measure: Number; unit: Participants
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Number analyzed (Participants) | 198 | 170 | 72 | 12
Participants
  AngioJet Thrombectomy without Lytic | 70 | 78 | 68 | 6
  AngioJet Thrombectomy + Lytic Delivery | 121 | 144 | 4 | 8
  Balloon Angioplasty | 144 | 120 | 59 | 4
  Stent Placement | 96 | 48 | 30 | 3
  Atherectomy | 8 | 0 | 0 | 0
  Filter Placement | 8 | 34 | 0 | 6
  Catheter Directed Thrombolysis | 76 | 79 | 1 | 3
  Non AngioJet Thrombectomy | 11 | 6 | 3 | 0

ADVERSE EVENTS:
Time Frame: Index procedure thru Discharge, 3 Month Follow Up
Description: Events that were related to initial index procedure and/or AngioJet.
Arm/Group | Limb Ischemia | Deep Vein Thrombosis | Hemodialysis Access | Other Thrombotic Conditions
Serious Adverse Events (participants affected / at risk) | 6/198 | 2/170 | 0/72 | 0/12
Other Adverse Events (participants affected / at risk) | 0/198 | 0/170 | 0/72 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Limb Ischemia (N=198) | Deep Vein Thrombosis (N=170) | Hemodialysis Access (N=72) | Other Thrombotic Conditions (N=12)
Bleeding Requiring transfusion (Surgical and medical procedures) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Renal Failure (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hemolytic Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Elevated Creatinine (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Non randomized observational registry

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days